CLINICAL TRIAL: NCT01433315
Title: Physiologic Effects of Sleep Restriction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Virend Somers, MD, PhD, MD, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 11-002121
Record Dates: First submitted 2011-08-15; First posted 2011-09-13 (Estimated); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Sleep Deprivation
Keywords: sleep deprivation; sleep restriction
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- sleep restriction (Experimental): restricted sleep during the experimental period
  Interventions: Behavioral: sleep restriction
- normal sleep (No Intervention): normal sleep during the experimental period

INTERVENTIONS:
Behavioral: sleep restriction — restricted sleep
  Arms: sleep restriction

SUMMARY:
Evidence suggests a relationship between sleep deprivation and cardiovascular disease. The investigators wish to determine whether 9 nights of modest sleep restriction results in activation of cardiovascular disease mechanisms, thus potentially increasing the risk of cardiovascular disease. The investigators hypothesize that sleep restriction will result in elevated blood pressure, inflammation, and neurocognitive deficits.

DETAILED DESCRIPTION:
Evidence suggests a relationship between sleep deprivation and cardiovascular disease. Voluntary sleep restriction is common, with 28% of the US adult population reports getting 6 or fewer hours of sleep per night, and those who do are 24% more likely to have cardiovascular disease and have twice the risk of hypertension. Insufficient sleep may conceivably be one of the most common, and most preventable, cardiovascular risk factors. The investigators wish to determine whether 9 nights of modest sleep restriction results in activation of cardiovascular disease mechanisms, thus potentially increasing the risk of cardiovascular disease. The investigators will combine our cardiovascular studies with state-of-the art sleep monitoring and neurocognitive tests to provide unambiguous data on the physiologic effects of sleep restriction. Together, the investigators findings will help explain whether the reduced sleep duration in the general population may be contributing to the current epidemic of cardiovascular disease, and suggest strategies to reduce this risk.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years
* No chronic medical conditions other than seasonal or environmental allergies
* On no prescription medications other than second generation antihistamines (Cetirizine, Fexofenadine, Desloratadine, Loratadine, etc), oral contraceptive pills, or intrauterine devices.
* BMI 18.5-35 kg/m2
* Both normotensive and prehypertensive people are eligible and will be studied
* Not a current smoker or tobacco user
* Not pregnant or breast feeding and not intending to become pregnant or breast feed

Exclusion Criteria:

* The investigators will exclude subjects who have any medical or psychiatric disorders
* History of anxiety or depression, and those taking any medications other than non-sedating antihistamines or oral contraceptives.
* Those found to have depression on a depression screening tool (BDI-II) will be excluded. Current smokers will be excluded.
* All female subjects will undergoing a screening pregnancy test and excluded if positive.
* Subjects found to have significant sleep disorders will be excluded.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2011-10; Primary Completion 2017-04-27 (Actual); Study Completion 2017-04-27 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure | throughout 16 days
  Change in mean arterial blood pressure over 24 hours, measured during acclimation, experimental, and recovery timepoints over the study period.

SECONDARY OUTCOMES:
Change in catecholamines | throughout 16 days
  Change in catecholamines, measured during acclimation, experimental, and recovery
Change in endothelial function | throughout 16 days
  Change in endothelial function, measured during acclimation, experimental, and recovery timepoints.
Change in baroreflex sensitivity | throughout 16 days
  Change in baroreflex sensitivity, measured during acclimation, experimental, and recovery
Change in arterial stiffness | throughout 16 days
  Change in arterial stiffness, measured during acclimation, experimental, and recovery timepoints.
Change in electrocardiographic characteristics | throughout 16 days
  Change in electrocardiographic characteristics, measured during acclimation, experimental, and recovery timepoints.
Change in markers of inflammation | throughout 16 days
  Change in markers of inflammation, measured during acclimation, experimental, and recovery timepoints.
Change in fat tissue characteristics | throughout 16 days
  Change in fat tissue characteristics, determined by analysis of a fat biopsy sample.

OTHER OUTCOMES:
Change in sleep architecture and sleepiness | throughout 16 days
  Change in sleep architecture and sleepiness, measured during acclimation, experimental, and recovery timepoints.
Change in neurocognitive function | throughout 16 days
  Change in neurocognitive function, measured during acclimation, experimental, and recovery timepoints
Change in cardiovascular reactivity | throughout 16 days
  Change in cardiovascular reactivity, measured during acclimation, experimental, and recovery timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Virend K Somers, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials